CLINICAL TRIAL: NCT00434941
Title: Multicenter Phase IV.II Trial, for the Administration of Capecitabine Simultaneous to Radiotherapy for Local Relapse Breast Cancer Patients With Negative Her2 Tumours
Brief Title: Capecitabine Plus Radiotherapy for Local Relapse Breast Cancer With Negative Her2 Tumours
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the slow rate of recruitment the study was stopped.
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2005-01
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Administration of capecitabine concomitant to radiotherapy; Her2: negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Radiotherapy

ARMS (1):
- Radiotherapy + Capecitabine (Experimental): Radiotherapy (for 25 days; Dose: 50 Gy) + Capecitabine (for 35 days; Dose: 825 mg/m2 twice per day p.o.) Experimental treatment consists of administration of 825 mg/m2 x 2 daily p.o., for 7 days simultaneously with daily radiotherapy treatment.Capecitabine will be administered for 35 days as maximum.
  Interventions: Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine
  Other Names: Xeloda
Radiation: Radiotherapy

SUMMARY:
This is a prospective, open-label, multicenter phase IV.II study. Patients with local relapse breast cancer will receive radiotherapy concomitant to the administration of capecitabine.

DETAILED DESCRIPTION:
Total dose of radiotherapy will be 50 Gy administered in daily session of 200 centigray (cGy). Radiotherapy treatment will not be longer than 6 weeks.

All patients will receive 1650 mg/m2 by mouth, per day (825 mg/m2 twice a day (p.o. bid) for 35 days.

Tissue samples must be analysed to determinate the human epidermal growth factor receptor-2 (HER2) by fluorescent in situ hybridization (FISH) technical.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histological diagnoses of operable invasive adenocarcinoma of the breast.
* Patients with tumour HER2 negative.
* Previous mastectomy surgery.
* Actual diagnoses of local recurrence of breast cancer.
* Patients must not present evidence of metastatic disease.
* Age >= 18 years old.
* Performance status (Karnofsky index) >= 70.
* Laboratory results (within 14 days prior to randomization):
* Hematology:

  * neutrophils >= 1.5 x 10e9/l;
  * platelets >= 100x 10e9/l;
  * hemoglobin >= 10 mg/dl
* Hepatic function:

  * total bilirubin <= 1,5 upper normal limit (UNL);
  * Alanine transaminase (SGOT) and aspartate aminotransferase (SGPT) <= 1.5 UNL;
  * alkaline phosphatase <= 1.5 UNL.
* Renal Function:

  * creatinine <= 175 µmol/l (2 mg/dl)or creatinine clearance >= 60 ml/min.

Exclusion Criteria:

* Distant metastasis or metastatic disease in organs.
* Metastasis in internal mammary chain lymph nodes
* Previous radiation treatment on the breast or other locations (30% or greater of the bone marrow).
* Prior treatment with continuous (greater than 24h) 5-fluorouracil (5-FU) infusion, capecitabine or other oral fluoropyrimidines such as eniluracil/5-FU , uracil/tegafur, S1 or emitefur.
* Known hypersensitivity to capecitabine, doxifluridine or any of its components.
* Organ allografts that require an immunosuppressor therapy.
* History of neurological or psychiatric disorders, which could preclude the patients to free informed consent.
* Clinically significant cardiac disease such as congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not well controlled with medication or history of myocardial infarction within the last 12 months or uncontrolled hypertension.
* Evidence of central nervous system (CNS) metastases. Pts with a history of uncontrolled seizures, CNS disorders or psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance should be excluded from the study.
* Pregnant or lactating women. Adequate contraceptive methods must be used during chemotherapy and hormone therapy treatments. Negative pregnancy test in the 14 previous days to randomization.
* Active uncontrolled infection or other severe pathologies such as active peptic ulcer, unstable diabetes mellitus.
* Major surgery during 4 weeks prior to treatment.
* Patients lacking physical integrity of upper gastrointestinal tract or with history of bad absorption syndrome.
* Anticoagulant treatment with coumadin anticoagulants.
* Concomitant treatment with other investigational products. Participation in other clinical trials with a non-marketed drug in the 30 previous days before randomization.
* Concomitant treatment with other therapy for cancer.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Complete clinical response rate | 28 days after the end of the radiotherapy
  The disease evaluation will be measured by RECIST criteria in the 28 days after the end of the radiotherapy by Magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Evaluation of the concomitant administration of capecitabine and radiotherapy as the first treatment | 28 days after the end of the radiotherapy
  Safety will be assessed by standard clinical and laboratory tests. Adverse events grade will be defined by the National Cancer Institute Common Terminology Criteria for Adverse (NCI-CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Clínico Universitario San Carlos
Locations (7):
- Spain (7):
  - Hospital Infanta Cristina, Badajoz
  - Hospital de la Esperanza, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- See also: Sponsor's website — http://www.geicam.org